CLINICAL TRIAL: NCT05925959
Title: Preoperative Weight Loss for Open Abdominal Wall Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin T. Miller (Other)
Responsible Party: Sponsor-Investigator, Benjamin T. Miller, Assistant Professor, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-418
Record Dates: First submitted 2023-06-14; First posted 2023-06-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Wall Hernia
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor of the patient reported outcomes will be blinded. Hernia recurrence will be assessed by blinded review of CT scans by 3 surgeons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront Surgery (No Intervention)
- Preoperative Weight Management Program (Active Comparator)
  Interventions: Other: Preoperative Weight Management Program

INTERVENTIONS:
Other: Preoperative Weight Management Program — The medical obesity intervention is comprised of monthly visits with an obesity medicine (OM) provider +/- a registered dietitian (in person or virtual). Lifestyle modifications (nutrition, physical activity, stress, sleep), appetite control, and medication side effects will be addressed in all visits. At initial visit, patients will evaluated in person by an OM provider +/- registered dietitian. An individualized intense lifestyle intervention will be implemented with the addition of an anti-obesity medication (phentermine, naltrexone/bupropion, phentermine/topiramate, liraglutide, semaglutide, etc). Medication use will be based on disease risk, patient preference, severity of obesity, contraindications, potential drug interactions and insurance coverage. A diet recommendation will be tailored to the patient's medical and food allergy history. Weight and vital signs will be monitored at each visit. Participants will have a total of 5 follow-up monthly encounters, every 30 +/- 7 days.
  Arms: Preoperative Weight Management Program

SUMMARY:
The goal of this randomized controlled trial is to compare preoperative intensive weight management to upfront surgery in obese patients undergoing complex abdominal wall reconstruction. The main question is will abdominal wall specific quality of life (using the HerQLes survey) for the group undergoing upfront surgery be non-inferior compared to the group in the weight management program.

DETAILED DESCRIPTION:
This is a prospective, single-center, registry-based, parallel, randomized controlled trial with 1:1 allocation. The study will consist of 2 arms: an intensive 6-month medical weight loss program prior to open retromuscular ventral hernia repair compared to upfront surgery without required weight loss. The medical obesity intervention will be conducted by physicians, nurse practitioners, and dieticians specializing in weight loss medicine. The study operations will be performed at Cleveland Clinic by six hernia surgeons with advanced abdominal wall reconstruction training.

ELIGIBILITY:
Inclusion criteria

* Adults having open retromuscular ventral hernia repair with an anticipated posterior component separation with transversus abdominis release and synthetic mesh
* BMI 40-55 kg/m2 and who are not planning to pursue weight loss surgery for any of the following reasons: they are not a candidate for weight loss surgery, cannot pursue weight loss surgery for insurance reasons, or are not interested in pursuing weight loss surgery.

Exclusion criteria

* Lack of English language fluency
* Urgent need for repair as determined by surgeon judgement
* Pregnant patients
* Permanent stoma in place
* Isolated flank hernia
* Anticipated need for staged operation; for example, patients who will undergo a mesh excision separate from definitive reconstruction.
* BMI <40 or >55 kg/m2
* Inability to participate in the Obesity Management Program due to lack of insurance coverage or history of mental illness (including eating disorders, schizophrenia, etc.).
* Obstructive symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal core health-specific quality of life at 1 year | 1 year
  This will be measured at 1 year using the HerQLes survey which is scored from 0-100 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Hernia recurrence at 1 year | 1 year
  This will be based on based on the current consensus definition of hernia recurrence which considers CT scan reviewed by 3 blinded assessors, surgeon clinical exam, and patient-reported bulge.
Wound morbidity at 30 days | 30 days
  This includes including surgical site infection, surgical site occurrence, and surgical site occurrence requiring procedural intervention.
Wound morbidity at 1 year | 1 year
  This includes including surgical site infection, surgical site occurrence, and surgical site occurrence requiring procedural intervention.
Body composition changes in weight | 1 year
  This includes comparative mean changes in body weight (kg) between groups from time of enrollment, day of surgery, 30-day follow-up, and 1-year follow-up.
Body composition changes in BMI | 1 year
  This includes comparative mean changes in BMI (kg/m2) between groups from time of enrollment, day of surgery, 30-day follow-up, and 1-year follow-up.
Patient abdominal wall specific- quality of life with preoperative weight management program | 1 year
  This includes difference in abdominal wall-specific quality of life using the HerQLes score (0-100 with higher scores indicating better abdominal wall-specific quality of life) in the weight loss arm before and after weight loss intervention.
Patient-reported pain changes with preoperative weight management program | 1 year
  This includes difference in pain using the PROMIS 3a Pain Intensity Score (30.7-71.8 with higher scores indicating more pain) in the weight loss arm before and after weight loss intervention.
Patient-reported quality of life changes with preoperative weight management program | 1 year
  This includes difference in overall quality of life using the EQ5D-5L with VAS (scored with an index value and a 0-100 score with higher scores indicating better quality of life) in the weight loss arm before and after weight loss intervention.
Abdominal wall -specific quality of life short-term | 30 days
  This includes difference in abdominal wall -specific quality of life using the HerQLes score between groups at baseline and 30 days postoperatively.
Pain scores | 1 year
  This includes the difference in pain scores using the PROMIS 3a Pain Intensity Score (scored from 30.7-71.8) at baseline, 30-day, and 1 year.
Cost effective analysis | 1 year
  Perform a formal cost effectiveness analysis.
Body weight percentage loss | 1 year
  Proportion of patients achieving a reduction in 5% and 10% body weight at end of 6-month medical weight loss intervention, day of surgery, and 1-year follow-up
Weight management program adherence | 1 year
  Proportion of successful completion of the program (defined as attending at least 4 visits) is associated with lower wound complications, hernia recurrence, or higher HerQLes score at one year
Impact of 10% body weight loss on wound complications | 1 year
  For patients with weight loss of 10% body weight prior to surgery compared to no weight loss prior to surgery - compare proportion of wound complications
Impact of 10% body weight loss on hernia recurrence | 1 year
  For patients with weight loss of 10% body weight prior to surgery compared to no weight loss prior to surgery - compare hernia recurrence at one year
Impact of 10% body weight loss | 1 year
  For patients with weight loss of 10% body weight prior to surgery compared to no weight loss prior to surgery - compare HerQLes score (0-100 with higher scores indicating better abdominal wall specific- quality of life) at one year
Urgent repair | 1 year
  Number of patients who require urgent hernia repair in either arm
Bariatric surgery prior to hernia repair and wounds | 1 year
  Number of patients who opt for bariatric surgery and, for those patients that undergo hernia repair, to evaluate rates of wound complications at one year
Bariatric surgery prior to hernia repair and hernia recurrence | 1 year
  Number of patients who opt for bariatric surgery and, for those patients that undergo hernia repair, to evaluate rates of hernia recurrence at one year
Bariatric surgery prior to hernia repair and abdominal wall specific quality of life | 1 year
  Number of patients who opt for bariatric surgery and, for those patients that undergo hernia repair and HerQLes scores (0-100 with higher scores indicating better abdominal wall specific- quality of life) at one year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Miller, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Remulla D, Miles KS, Carvalho A, Maskal SM, Butsch WS, Beffa LR, Petro CC, Krpata DM, Prabhu AS, Rosen MJ, Miller BT. Preoperative weight loss for open abdominal wall reconstruction: study protocol for a randomized controlled trial. Hernia. 2025 May 28;29(1):187. doi: 10.1007/s10029-025-03375-y. PMID 40434485